CLINICAL TRIAL: NCT01721824
Title: IPS-MA - A Randomized Clinical Trial Examining the Effect of a Modified IPS Intervention in Addition to Treatment as Usual Versus Treatment as Usual Alone for Individuals With Mood or Anxiety Disorders
Brief Title: The Effect of IPS-MA- A Modified Early Supported Employment Intervention for Individuals With Mood or Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-2-2011-FSP20
Record Dates: First submitted 2012-10-24; First posted 2012-11-06 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Affective Disorder; Major Depressive Disorder; Bipolar Disorder; Anxiety Disorder
Keywords: Supported employment; Individual Placement and Support; Workability; Return to work
MeSH Terms: conditions — Mood Disorders; Depressive Disorder, Major; Bipolar Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPS-MA (Experimental): The IPS-MA method consists of five basic services for the participants. 1)Individual mentor support, based on psychiatric knowledge. 2)Coordination by the mentor of activities, internal as well as from external providers. 3)Career counseling aimed at people with mental illnesses. 4)Impartial help to clarify private economy. 5) Contact to employers to help participants obtain jobs, and keep them.
  Participants will receive the IPS-MA method in addition to treatment as usual.
  Interventions: Behavioral: The IPS-MA method
- Control group (No Intervention): Participants randomised to the control group will receive "treatment as usual" only. This means the standard support offered by the social- and health services in Denmark.

INTERVENTIONS:
Behavioral: The IPS-MA method — During the first 6 months participants are usually offered 3 meetings with their mentor per month, lasting approximately 1 1/2 hours each. The following 6 months they are offered 1 meeting per month, lasting approximately 1 hour. The estimated duration of the IPS-MA intervention is 12 months, but since the needs of the participants are very individual, this may vary.
  Other Names: IPS-modified for people recently diagnosed with mood or anxiety disorders (IPS-MA)
  Arms: IPS-MA

SUMMARY:
The aim of the present study, is to evaluate the effect of a supported employment intervention, IPS-modified for people with mood and anxiety (IPS-MA) on employment or education, when offered to people with onset mood or anxiety disorders who are not likely to be able to return to work within three month.

The hypothesis is that the IPS-MA method is associated with a shorter recovery period and more people returning to work or education, compared to treatment as usual.

DETAILED DESCRIPTION:
Background: The IPS-MA method is a modified Individual Placement and Support (IPS) intervention, aiming at supporting people with mood or anxiety disorders regain their workability and return to work or education. Previous studies have showed, that IPS has an effect on employment when offered to people with severe mental illness. Further studies are crucial to demonstrate whether the modified IPS, the IPS-MA method, has an effect when offered to people with mood or anxiety disorders who are not yet chronified.

Methods/design:The trial design is a randomized, assessor-blinded, clinical trial of the IPS-MA method in addition to treatment as usual compared to treatment as usual alone for 326 participants diagnosed with a mood or anxiety disorder, living in the Capital Region of Denmark. The primary outcome is competitive employment or education. Secondary outcomes are days of competitive employment or education, disease symptoms, level of functioning, and quality of life at follow-up 12 and 24 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed following the International Classification of Diseases (ICD-10) criteria of affective disorder (F30-39) or anxiety disorder (F40-41)
* Not able to work within 3 months
* Associated with the Mental Health Center Copenhagen, Frederiksberg, Hillerød, Hvidovre or Ballerup
* Only having had contact to the Mental Health services during the past 3 years
* Having had competitive employment or attending a study within the past two years.
* Has returning to work or education as an important goal
* Under the age of 60
* Able to speak, read and understand danish
* Has given informed consent verbally and in writing

Exclusion Criteria:

* A somatic disease that effects the workability
* Substance og alcohol abuse
* have a guardian or a forensic psychiatric arrangement
* not given informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2011-10; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Competitive employment or education | 24 months
  Competitive employment includes being on rehabilitation benefits, flexible jobs and wage subsidy job. Information on employment and education will be extracted from the DREAM database. This database is administered by The National Labour Market Authority and contains information on employment, sickness leave, educations eligible to state education grant, pre-vocational training, disability pension, social security, and sickness benefits.

SECONDARY OUTCOMES:
Number of days of competitive employment or studying | 24 months
  Information will be obtained from the Dream database.
Hamilton Rating Scale for Depression - 6 items | 24 months
  Level of symptoms of depression
Hamilton Rating Scale for anxiety -6 item scale | 24 months
  Level of symptoms of anxiety
Global Assessment of Function (GAF-F) | 24 months
  Level of function
WHO-5 well-being index | 24 months
  Level of health-related quality of life

OTHER OUTCOMES:
Competitive employment or studying | 12 months
  Competitive employment includes being on rehabilitation benefits, flexible jobs and wage subsidy jobs. Information on employment and education will be extracted from the DREAM database. The database is administered by The National Labour Market Authority and contains information on employment, sickness leave, educations eligible to state education grant, pre-vocational training, disability pension, social security, and sickness benefits.
Changing from matchgroup 2 or 3 to matchgroup 1 | 12 and 24 months
  If participants are matchgroup 2 or 3, they are not able to go back to work within the following 3 months. If participants are matchgroup 1, they should be actively seeking jobs.
Number of days of competitive employment or studying | 12 and 24 months
  Information will be obtained from the Dream database.
Time until returning to employment or education | 24 months
  Information will be obtained from the Dream database.
Hamilton Rating Scale for Depression - 6 items | 12 months
  Level of symptoms of depression
Hamilton Rating Scale for anxiety -6 item scale | 12 months
  Level of symptoms of anxiety
The Bech-Rafaelsen Mania Scale (MAS) | 12 and 24 months
  Level of symptoms af mania
Global Assessment of Function (GAF-F) | 12 months
  Level of function
Personal and Social Performance (PSP) | 12 and 24 months
  Social performance in four domains (socailly usefull activities, personal and social relationships, self-care and disturbing and aggressive behaviour)
WHO-5 well-being index | 12 months
  Level of health-related quality of life
Sheehan Disability Scale (SDS) | 12 and 24 months
  Level of function regarding social relationships, work, spare time and family.
The Empowerment Scale | 12 and 24 months
The Changes Questionnaire | 12 and 24 months
  Motivation to seeking employment or education
The Client Satisfaction Questionnaire | 12 and 24 months
  Satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, MD, PhD, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Mental Health Center Ballerup, Mental Health Center Frederiksberg, Mental Health Center Copenhagen, and Mental Health Center of Northern Seeland, Ballerup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell K, Bond GR, Drake RE. Who benefits from supported employment: a meta-analytic study. Schizophr Bull. 2011 Mar;37(2):370-80. doi: 10.1093/schbul/sbp066. Epub 2009 Aug 6. PMID 19661196
- [Background] Bond GR, Drake RE, Becker DR. An update on randomized controlled trials of evidence-based supported employment. Psychiatr Rehabil J. 2008 Spring;31(4):280-90. doi: 10.2975/31.4.2008.280.290. PMID 18407876
- [Derived] Hellstrom L, Christensen TN, Bojesen AB, Eplov LF. Predictors of Return to Work for People with Anxiety or Depression Participating in a Randomized Trial Investigating the Effect of a Supported Employment Intervention. J Occup Rehabil. 2023 Mar;33(1):61-70. doi: 10.1007/s10926-022-10046-7. Epub 2022 May 25. PMID 35612640
- [Derived] Hellstrom L, Madsen T, Nordentoft M, Eplov LF. Trajectories of symptoms of anxiety and depression among people on sick leave with mood or anxiety disorders: Secondary analysis from a randomized controlled trial. J Psychiatr Res. 2021 May;137:250-257. doi: 10.1016/j.jpsychires.2021.02.040. Epub 2021 Feb 25. PMID 33714077
- [Derived] Hellstrom L, Madsen T, Nordentoft M, Bech P, Eplov LF. Trajectories of Return to Work Among People on Sick Leave with Mood or Anxiety Disorders: Secondary Analysis from a Randomized Controlled Trial. J Occup Rehabil. 2018 Dec;28(4):666-677. doi: 10.1007/s10926-017-9750-x. PMID 29282650
- [Derived] Hellstrom L, Bech P, Hjorthoj C, Nordentoft M, Lindschou J, Eplov LF. Effect on return to work or education of Individual Placement and Support modified for people with mood and anxiety disorders: results of a randomised clinical trial. Occup Environ Med. 2017 Oct;74(10):717-725. doi: 10.1136/oemed-2016-104248. Epub 2017 May 25. PMID 28546319
- [Derived] Hellstrom L, Bech P, Nordentoft M, Lindschou J, Eplov LF. The effect of IPS-modified, an early intervention for people with mood and anxiety disorders: study protocol for a randomised clinical superiority trial. Trials. 2013 Dec 24;14:442. doi: 10.1186/1745-6215-14-442. PMID 24368060